CLINICAL TRIAL: NCT04628091
Title: Characterization of Persistent Organic Pollutants Exposure During Preconception and Preimplantation Development in the Human Fallopian Tube: TUBPOP.
Brief Title: Characterization of Persistent Organic Pollutants Exposure During Preconception and Preimplantation Development.
Acronym: TUBPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/19/0257; RC31/19/0257 (Other Grant/Funding Number: Biomedicine Agency)
Record Dates: First submitted 2020-11-06; First posted 2020-11-13 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Exposure to Environmental Pollution
Keywords: Chemical exposome; Fallopian tube; Persistent Organic Pollutants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): Test group is composed of 20 women of reproductive age devoid of any pathology coming to the hospital for a salpingectomy for contraceptive purposes or for a total hysterectomy.
  Interventions: Other: Sampling on surgery day

INTERVENTIONS:
Other: Sampling on surgery day — In the morning, the day of the surgery (the patient will be fasting):
  * Occipital hair sample (without roots)
  * Venous blood sample (3 tubes of 7mL)
  During the surgery:
  * Sample of 0.5 to 1 cm3 of subcutaneous adipose tissue during laparoscopic umbilical access
  * Collection of a portion of Ampulla proximal part and Isthmus distal part in order to obtain a piece of approximately 4 cm long (2cm of ampulla and 2 cm of isthmus) for each tube.

SUMMARY:
In order to evaluate if gametes and preimplantation embryos are in vivo exposed to environmental chemicals, the detection of 6 molecules representative of 3 persistent organic pollutants families will be performed in the mucosa of fallopian tubes obtained after bilateral salpingectomy performed for sterilization purpose in 20 women and compared with concentrations in adipose tissue. This feasibility study is a preliminary step before larger clinical surveys and in vitro studies.

DETAILED DESCRIPTION:
The fallopian tube is the physiological environment of the mature gametes and the preimplantation embryo. While animal and epidemiological data are accumulating that demonstrate the role of alterations of the fetal environment in the programming of post-natal development and health at adulthood, the impact of environmental perturbations during early development (fertilization and preimplantation development) is mainly shown by animal studies (apart persistent questions about health of children conceived after assisted reproductive technologies). Animal expositions to chemical contaminants of the environment targeted on the preimplantation period have been shown to alter health at adulthood. In the same way, in vitro short exposition of male or female gametes to some of these chemicals can impact their functions. It is therefore important to characterize the chemical environment of gametes and preimplantation embryo in the human fallopian tube.

This project aims to demonstrate the feasibility of quantitative measurements for 3 families of persistent environmental contaminants at the oviduct level. In women of reproductive age devoid of any pathology able to alter tubal mucosa, fallopian tubes will be recovered after laparoscopic bilateral salpingectomy performed with the goal of sterilization. Concentrations in the tubal mucosa tissue will be analyzed for at least 2 representative members of 3 chemicals families (organochlorine pesticides (DDE, HCB), polychlorobiphenyls (PCB 153 and 138) and flame retardants (PBDE47 and 153). A comparison with the concentration obtained in the adipose tissue collected at the time of umbilical incision for laparoscopy and in blood will allow to evidence the exposition of each women to each type of contaminant. One bundle of hair strand will be collected from the occipital region of the head and stored for further analysis.

This project is a feasibility study on 20 women but its perspectives are numerous. It is supported by a solid consortium that will assure the recruitment of the women in this indication and its technical implementation.

ELIGIBILITY:
Inclusion Criteria:

* Addressed to surgery for a voluntary sterilization purpose by bilateral salpingectomy or for total hysterectomy (due to pelvic organs prolapse, functional menorrhagia)
* No previous pathology affecting directly or indirectly the tubal mucosa
* Regular menstrual cycles (26 to 34 days) or under estro-progestative contraceptive
* National health insurance affiliation or equivalent
* Informed and free consent

Exclusion Criteria:

* Absence of 1 or 2 fallopian tubes
* Current or previous disease with persistent effect on tubal mucosa (salpingitis, hydrosalpinx, medically treated extra-uterine pregnancy)
* BRCA1 or 2 mutation in the subject or her first-degree relatives (parents, siblings, children)
* ovarian cancer before age of 50 in a first-degree relative
* uterine, tubal or ovarian anomaly visualized on a presurgical imagery and necessitating a total anatomopathological examination of one of the fallopian tube or a macroscopic anomaly visualized during surgery necessitating a total anatomopathological examination of one of the fallopian tube
* Contraception using progestative alone
* Ovarian desensitisation using gonadotropin-releasing hormone (GnRH) agonists
* Bariatric surgery in the previous year
* Placement under judicial protection, guardianship, or supervision

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects for whom a quantifiable detection for the 6 molecules is obtained | During surgery
  A proportion above or equal to 90 % (quantification in 18 women out of 20 at least) will be the threshold retained as a possible quantification.

SECONDARY OUTCOMES:
Comparison of intratubal and adipose tissue concentrations of the 6 toxicants | During surgery
  For each of the 6 toxicants, a comparison between the observed intratubal and adipose concentrations will be made within the population and a linear or non-linear relationship will be sought.

CONTACTS AND LOCATIONS:
Overall Officials: Roger LEANDRI, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rappaport SM. Genetic Factors Are Not the Major Causes of Chronic Diseases. PLoS One. 2016 Apr 22;11(4):e0154387. doi: 10.1371/journal.pone.0154387. eCollection 2016. PMID 27105432
- [Background] Lee DH, Jacobs DR Jr, Porta M. Hypothesis: a unifying mechanism for nutrition and chemicals as lifelong modulators of DNA hypomethylation. Environ Health Perspect. 2009 Dec;117(12):1799-802. doi: 10.1289/ehp.0900741. Epub 2009 Jul 8. PMID 20049195
- [Background] Dereumeaux C, Saoudi A, Pecheux M, Berat B, de Crouy-Chanel P, Zaros C, Brunel S, Delamaire C, le Tertre A, Lefranc A, Vandentorren S, Guldner L. Biomarkers of exposure to environmental contaminants in French pregnant women from the Elfe cohort in 2011. Environ Int. 2016 Dec;97:56-67. doi: 10.1016/j.envint.2016.10.013. Epub 2016 Oct 24. PMID 27788374
- [Background] Lee WC, Fisher M, Davis K, Arbuckle TE, Sinha SK. Identification of chemical mixtures to which Canadian pregnant women are exposed: The MIREC Study. Environ Int. 2017 Feb;99:321-330. doi: 10.1016/j.envint.2016.12.015. Epub 2016 Dec 29. PMID 28040263
- [Background] Watkins AJ, Fleming TP. Blastocyst environment and its influence on offspring cardiovascular health: the heart of the matter. J Anat. 2009 Jul;215(1):52-9. doi: 10.1111/j.1469-7580.2008.01033.x. Epub 2009 Feb 9. PMID 19215321